CLINICAL TRIAL: NCT01911741
Title: A Phase I, Single-center, Open-label, Randomized, Parallel, Relative Bioavailability Study Comparing a Capsule and Tablet Formulations of Enzalutamide Following a Single 160 mg Dose Under Fasted Conditions in Healthy Male Subjects
Brief Title: A Study to Compare Capsule and Tablet Forms of MDV3100 (Enzalutamide) After Administration of a Single Set Dose Under Fasted Conditions in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 9785-CL-0010; 2012-002502-49 (EudraCT Number)
Record Dates: First submitted 2013-07-26; First posted 2013-07-30 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Healthy Subjects; Castration Resistant Prostate Cancer (CRPC); Relative Bioavailability; MDV3100
Keywords: Phase I; Enzalutamide; Relative bioavailability of MDV3100; Immediate release oral formulation; Xtandi
MeSH Terms: interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental): Single dose of 4 liquid-filled capsules of MDV3100 reference formulation
  Interventions: Drug: MDV3100
- Treatment B (Experimental): Single dose of 2 tablets of MDV3100 formulation tablet B
  Interventions: Drug: MDV3100
- Treatment C (Experimental): Single dose of 2 tablets of MDV3100 formulation tablet C
  Interventions: Drug: MDV3100

INTERVENTIONS:
Drug: MDV3100 — Oral
  Other Names: enzalutamide; Xtandi

SUMMARY:
A study to evaluate the bioavailability (BA) of a single oral dose of MDV3100 (enzalutamide) formulated as a solid spray dried tablet compared to oral liquid-filled capsules, and the safety and tolerability of oral formulations.

Subjects are admitted to the clinic from days 1 to 5, followed by outpatient assessments up to Day 50. They return to the clinic for an end of study visit (ESV) 7-10 days after the last pharmacokinetic (PK) sampling or after early withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a body mass index (BMI) range of 18.5 - 29.9 kg/m2, inclusive. The subject weighs at least 50 kg (screening).
* Male subject and his female spouse/partner who is of childbearing potential must be using highly effective contraception consisting of two forms of birth control (one of which must be a barrier method) starting at screening and continue throughout the study period and for 3 months after final study drug administration.
* Male subject must not donate sperm starting at screening and throughout the study period and for at least 3 months after final study drug administration.

Exclusion Criteria:

* Known or suspected hypersensitivity to enzalutamide, or any components of the formulation used.
* Confirmed CYP2C8 poor metabolizer status based on genotyping analysis.
* Any history of seizure including a febrile seizure in childhood, loss of consciousness, transient ischemic attack, or any condition that may pre-dispose to seizure.
* The subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection), or fungal (non-cutaneous) infection within 1 week prior to first clinic check in.
* Use of grapefruit or marmalade in the week prior to admission to the Clinical Unit, as reported by the subject.
* Any significant blood loss, donated one unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to clinic admission on Day -1.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2012-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Relative BA of capsule and tablet formulations of enzalutamide following a single dose of enzalutamide under fasted conditions | Day 1 through Day 50 (26 times)
  AUC0-t (Area Under Curve from time zero to last quantifiable sample), AUC0-inf (AUC extrapolated to infinity), Cmax (Maximum concentration)

SECONDARY OUTCOMES:
Relative BA of capsule and tablet formulations of enzalutamide following a single dose of enzalutamide under fasted conditions | Day 1 through Day 50 (26 times)
  AUC0-72h (AUC from time zero to 72h post dose), AUC0-t, AUC0-inf, %AUC (Percentage of AUC), Cmax, tmax (Time to attain Cmax), λz (Terminal elimination rate constant), t1/2 (Terminal elimination half life), (MPR) metabolites to parent ratio, MPR(molecular weight corrected [MWC]), %AUC, CL/F (apparent oral clearance), Vz/F (apparent volume of distribution)
Safety and tolerability of oral formulations of enzalutamide | Screening through ESV (7-10 days after the last pharmacokinetic (PK) sampling or after early withdrawal)
  adverse events, physical examination, vital signs, clinical laboratory tests, 12-lead Electrocardiogram (ECG)

CONTACTS AND LOCATIONS:
Overall Officials: Study Manager, Study Chair — Astellas Pharma Europe B.V.
Locations (1):
- Parexel International GmbH, Berlin, Germany